CLINICAL TRIAL: NCT03682549
Title: Oral Microbiome of Patients With Chronic Hepatitis C Virus Infection: A Case-Control Study
Brief Title: Oral Microbiome of Patients With Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, Principal investigator, Cairo University
Other Study IDs: A1PhD
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis C Viral
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A Swab from the buccal mucosa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCV positive Patients: patients will be recruited from the outpatient's viral hepatitis clinic
  The patients will be diagnosed as HCV positive through (antiHCV-Ab) and (HCV-PCR) tests
  Interventions: Diagnostic Test: Oral microbiome analysis
- Successfully treated former HCV patients: Patients formerly diagnosed as HCV positive who received DAA treatment successfully.
  Interventions: Diagnostic Test: Oral microbiome analysis
- Normal Individuals: healthy volunteers recruited from the outpatient clinic of the Faculty of Dentistry- Cairo University
  Interventions: Diagnostic Test: Oral microbiome analysis

INTERVENTIONS:
Diagnostic Test: Oral microbiome analysis — Oral swab from the buccal mucosa will be obtained and then analysed Oral Microbiome analysis:The microbial RNA will be sequenced using Next Generation Sequencer.

SUMMARY:
Hepatitis C virus (HCV) infection is very common in Egypt and the middle east. The disease affects multiple body organs and may proceed to hepatocellular carcinoma. The viral disease causes changes in the microbial symbiosis in the human body. Thus, the analysis of the microbiome may provide a means of diagnosis for HCV infection.

Thus, this study will be held to detect if the microbiome of patients having HCV differ from that of normal individuals.

DETAILED DESCRIPTION:
Human oral cavity is a great habitat for more than 600 species of bacteria, known as oral microbiota, living in equilibrium. Oral microbiota plays an important role in maintaining oral health; however when the balance in oral bacterial population is disturbed- known as dysbiosis- oral and systemic diseases may arise.

Some systemic diseases were proven to be associated with oral dysbiosis. Among these diseases are diabetes mellitus, cardiovascular diseases, breast cancer, pancreatic cancer, autoimmune liver diseases, hepatic encephalopathy and hepatitis B infection.

Hepatitis C virus (HCV) is considered an epidemic disease in Egypt; affecting about 10% of Egyptians ranging between 15 and 59 years of age. HCV infection damages the liver progressively causing liver cirrhosis, hepatic encephalopathy and may proceed to hepatocellular carcinoma.

Due to being a serious disease, together with the promising results of the newly discovered directly acting antiviral agents in treatment of chronic HCV, medicine has been concerned with finding efficient methods for its early diagnosis; in order to ensure early effective treatment and prevent serious complications.

Evidence suggests that a link exists between dysbiotic oral microenvironment and liver disease through oral-liver-gut axis. Attempts have been made to investigate the complex oral microbiota. With the advent of whole-genome sequencing technology, the genome of microbes have been possible to be sequenced in what is known as microbiome. Analyzing the genome of complex environment containing multiple individual microbes is called metagenomics.

Oral microbiome depends on sequencing of the 16S rRNA to provide a map of all oral microbiota available in the oral cavity. The technology of oral microbiome sequencing advanced from Sanger sequencing, that had shallow sequencing effort, to high throughput sequencing combined with bioinformatic tools, that allowed for comprehensive study of the complex microbiome.

Dysbiosis has been used for diagnosis of liver diseases through stool analysis. Only one study used oral dysbiosis to diagnose hepatic encephalopathy and another one used it in testing hepatitis B infection. However, oral dysbiosis has not been used to diagnose HCV infection before.

Understanding the oral microbiome at state of health and its change at state of disease can help predict the early stages of disease and treat it before further damage and disease progression occur. It can also help treat each patient according to the specific microbiome detected through personalized medicine. Furthermore, targeted treatment to each patient's specific microbiome can be introduced using specific prebiotics and probiotics to maintain the bacterial symbiosis and so assist the immune system in its continuous antiviral battle.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients 18 years or older. 2. Non-smokers

Exclusion Criteria:

* 1. Patients who took any antibiotic or probiotics in the past month. 2. Patients having known active bacterial, fungal or other viral disease. 3. Patients having clinically apparent oral disease. 4. Patients undergoing radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be divided into three groups:
  Group I: Patients diagnosed with Hepatitis C virus. Group II: successfully treated chronic HCV patients Group III: Healthy individuals
  They will be asked to rinse gently, then buccal mucosal swabbing takes place.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Oral Microbiome dysbiosis | 1 month
  changes in oral microbial composition will be analysed using bioinformatics tools to provide figures showing the extent of dysbiosis and its composition

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No